CLINICAL TRIAL: NCT01621633
Title: A Single-dose, Open-label Parallel-group Study to Assess the Pharmacokinetics of LCZ696 in Subjects With Hepatic Impairment Compared to Matched Healthy Subjects
Brief Title: A Study of LCZ696 in Subjects With Mild and Moderate Hepatic Impairment Compared With Normal Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CLCZ696B2203; 2012-000983-27 (EudraCT Number)
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-07

CONDITIONS: Hepatic Impairment
Keywords: hepatic impairment
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: mild hepatic impairment (Experimental): LCZ696 200 mg, given as a single oral dose
  Interventions: Drug: LCZ696
- Group 2: moderate hepatic impairment (Experimental): LCZ696 200 mg, given as a single oral dose
  Interventions: Drug: LCZ696
- Group 3: healthy volunteers (Experimental): LCZ696 200 mg, given as a single oral dose. Each healthy volunteer will match in race, age (±5 years), gender, weight (±15%) to an individual subject with hepatic impairment in groups 1 and 2
  Interventions: Drug: LCZ696

INTERVENTIONS:
Drug: LCZ696

SUMMARY:
This is a study to characterize the pharmacokinetics as well as safety and tolerability of a single oral dose of LCZ696 200 mg in subjects with mild and moderate hepatic impairment compared to matched healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* All subjects:

  * Male and female subjects aged 18-75 years.
  * Body weight at least 55 kg with a body mass index between 18-35 kg/m2.
* Hepatic impairment subjects:

  * Mild or moderate hepatic impairment.

Exclusion Criteria:

* All subjects:

  * Clinical manifestations of postural symptomatic hypotension at screening or baseline.
  * History of hypersensitivity to LCZ696 or to drugs of similar classes.
* Hepatic impairment subjects:

  * Hepatic impairment due to non-liver disease.
  * Treatment with any vasodilator, autonomic alpha blocker or beta2 agonist within 2 weeks of dosing.
  * Encephalopathyy Stage III or IV.
  * Primary biliary liver cirrhosis or biliary obstruction.
  * History of gastro-intestinal bleeding within 3 months prior to screening.
* Healthy subjects:

  * Any surgical or medical condition which might significantly alter the distribution, or excretion of drugs, or which may jeopardize the subject in case of participation in the study.
  * Use of prescription drugs, herbal supplements, and/or over-the-counter medication, dietary supplements (vitamins included) within 2 weeks prior to initial dosing.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Grünstadt, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants received the study treatment according to the population subset that was defined based on the severity of hepatic impairment and healthy volunteers: Group 1, subjects with mild hepatic impairment; Group 2, subjects with moderate hepatic impairment; Groups 3 and 4, healthy volunteers matching to Groups 1 and 2, respectively.
Groups:
- Participants With Mild Hepatic Impairment (HI); Participants With Moderate Hepatic Impairment (HI): LCZ696 200 mg, given as a single oral dose
- Healthy Volunteers (Mild HI Matched): LCZ696 200 mg, given as a single oral dose. Each healthy volunteer matched in race, age (±5 years), gender, weight (±15%) to an individual subject with hepatic impairment in group 1
- Healthy Volunteers (Moderate HI Matched): LCZ696 200 mg, given as a single oral dose. Each healthy volunteer matched in race, age (±5 years), gender, weight (±15%) to an individual subject with hepatic impairment in group 2
Period: Overall Study
Arm/Group | Participants With Mild Hepatic Impairment (HI) | Participants With Moderate Hepatic Impairment (HI) | Healthy Volunteers (Mild HI Matched) | Healthy Volunteers (Moderate HI Matched)
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Mild Hepatic Impairment (HI) | Participants With Moderate Hepatic Impairment (HI) | Healthy Volunteers (Mild HI Matched) | Healthy Volunteers (Moderate HI Matched) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.1 (7.92) | 57.9 (11.67) | 58.9 (8.68) | 60.3 (11.21) | 59.0 (9.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 1 | 8
  Male | 5 | 7 | 5 | 7 | 24

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of LCZ696 Analytes (AHU377, LBQ657, and Valsartan)
Description: Blood samples were taken on Day 1 (treatment day) within 60 minutes prior to dosing, then, 0.5,1,1.5,2,3,4,6,8,12 hours after the dosing and on Days 2, 3, 4 and 5 post dosing
Time Frame: From pre-dose on Day 1 until 96h post-dose (Day 5)
Population: PK analysis set: The PK analysis set included all subjects with at least one available, valid (i.e. not flagged for exclusion) PK concentration measurement, who received any study drug, and experienced no protocol deviations with relevant impact on PK data.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Participants With Mild Hepatic Impairment (HI) | Participants With Moderate Hepatic Impairment (HI) | Healthy Volunteers (Mild HI Matched) | Healthy Volunteers (Moderate HI Matched)
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng*hr/mL
  AHU377 | 2540 (1010) | 6200 (2970) | 1580 (390) | 1740 (520)
  LBQ657 | 118000 (37000) | 173000 (99900) | 77900 (14700) | 83100 (14700)
  Valsartan | 28500 (16900) | 63800 (48700) | 21600 (5980) | 25300 (11800)

2. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero Extrapolated to Infinite Time [AUCinf)] of LCZ696 Analytes (AHU377, LBQ657, and Valsartan)
Description: as for outcome 1
Time Frame: From pre-dose on Day 1 until 96h post-dose (Day 5)
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Participants With Mild Hepatic Impairment (HI) | Participants With Moderate Hepatic Impairment (HI) | Healthy Volunteers (Mild HI Matched) | Healthy Volunteers (Moderate HI Matched)
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng*hr/mL
  AHU377 | 2540 (1010) | 6200 (2980) | 1590 (390) | 1740 (519)
  LBQ657 | 121000 (41000) | 187000 (124000) | 78500 (14700) | 84100 (14800)
  Valsartan | 28800 (16900) | 65600 (50100) | 21900 (5950) | 26500 (12400)

3. Primary Outcome: Maximum Plasma Concentration (Cmax) for LCZ696 Analytes (AHU377, LBQ657, and Valsartan)
Description: as for outcome 1
Time Frame: From pre-dose on Day 1 until 96h post-dose (Day 5)
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Participants With Mild Hepatic Impairment (HI) | Participants With Moderate Hepatic Impairment (HI) | Healthy Volunteers (Mild HI Matched) | Healthy Volunteers (Moderate HI Matched)
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL
  AHU377 | 2530 (1400) | 4430 (1760) | 1510 (585) | 1410 (445)
  LBQ657 | 7730 (1470) | 6690 (917) | 7450 (1320) | 6770 (1710)
  Valsartan | 4000 (2310) | 4180 (2340) | 3880 (1490) | 3730 (1540)

4. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Death
Description: Adverse events, serious adverse events and death were monitored from screening to end of study
Time Frame: From the screening visit until Day 5
Population: Safety set: The safety set includes all participants who received study treatment.
Measure: Number; unit: Participants
Arm/Group | Participants With Mild Hepatic Impairment (HI) | Participants With Moderate Hepatic Impairment (HI) | Healthy Volunteers (Mild HI Matched) | Healthy Volunteers (Moderate HI Matched)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Participants
  Adverse events (serious and non-serious) | 0 | 2 | 0 | 0
  Serious adverse events | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Moderate Hepatic Impaired Patients: Moderate hepatic impaired patients
Arm/Group | Moderate Hepatic Impaired Patients | Healthy Volunteers (Mild HI Matched) | Healthy Volunteers (Moderate HI Matched) | Participants With Mild Hepatic Impairment (HI)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 0/8 | 0/8 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate Hepatic Impaired Patients (N=8) | Healthy Volunteers (Mild HI Matched) (N=8) | Healthy Volunteers (Moderate HI Matched) (N=8) | Participants With Mild Hepatic Impairment (HI) (N=8)
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0
BLOOD POTASSIUM DECREASED (Investigations) | 1 | 0 | 0 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.